CLINICAL TRIAL: NCT07340229
Title: Effects of Laughter Yoga on Psychological Resilience and Coping Attitudes in Mothers of Children in the Pediatric Intensive Care Unit: A Randomized Controlled Trial
Brief Title: Effects of Laughter Yoga in Mothers of PICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Sadiye Dur, Associate Professor, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IDU-NURSING-SD-01
Record Dates: First submitted 2026-01-02; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Laughter Yoga
Keywords: Pediatric Intensive Care Unit; Resilience; Coping Skills; Family Centered Nursing; Laughter Therapy; Laughter
MeSH Terms: conditions — Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: A total of 40 mothers were randomly assigned to either the laughter yoga group (n = 20) or control group (n = 20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga Group (Experimental): Mothers in the intervention group participated in structured laughter yoga sessions lasting 15-20 minutes, conducted over a period of 3-4 days.
  Interventions: Behavioral: Laughter Yoga
- Control Group (No Intervention): The control group received routine care only.

INTERVENTIONS:
Behavioral: Laughter Yoga — Mothers in the intervention group participated in structured laughter yoga sessions lasting 15-20 minutes, conducted over a period of 3-4 days.
  Arms: Laughter Yoga Group

SUMMARY:
This randomized controlled trial examined the effects of laughter yoga on resilience and coping attitudes in mothers of children hospitalized in the pediatric intensive care unit. Mothers whose children had been hospitalized for at least one week were randomly assigned to an intervention or control group. The intervention group participated in structured laughter yoga sessions lasting 15-20 minutes over 3-4 days, while the control group received routine care. Psychological resilience and coping attitudes were assessed using standardized measurement tools. The study aimed to provide evidence for a brief, non-pharmacological intervention to support maternal psychological well-being in PICU settings.

DETAILED DESCRIPTION:
Having a child hospitalized in a pediatric intensive care unit (PICU) is a highly stressful experience for parents, particularly mothers, and is often associated with increased psychological distress, reduced resilience, and ineffective coping strategies. Despite the critical importance of supporting parental mental well-being in PICU settings, there is a lack of evidence-based, non-pharmacological interventions that simultaneously target resilience and coping attitudes.

This study aimed to evaluate the effect of laughter yoga on resilience and coping attitudes in mothers of children in the pediatric intensive care unit.

A single-blind, parallel-group randomized controlled trial was conducted with the mothers of children hospitalized in the PICU for at least one week. Mothers in the intervention group participated in structured laughter yoga sessions lasting 15-20 minutes over 3-4 days, while the control group received routine care only. Data were collected using the Connor-Davidson Resilience Scale and the Coping Attitudes Assessment Scale before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged 18 years or older
* Ability to read and speak Turkish
* Having a child hospitalized in the pediatric intensive care unit (PICU) for at least one week
* Access to basic communication tools (telephone and/or internet)
* No previous participation in laughter yoga or a similar intervention

Exclusion Criteria:

* Presence of a clinically diagnosed severe psychiatric disorder
* Having a child who was terminally ill or clinically unstable
* Participation deemed inappropriate by the attending physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale | Six months
  The Connor-Davidson Resilience Scale (CD-RISC-10) was originally developed by Connor and Davidson (2003), subsequently shortened to 10 items by Campbell-Sills and Stein (2007), and adapted to Turkish by Sarıçam (2010). The scale is scored using a five-point Likert-type format (0-4), with higher total scores indicating greater resilience. In the Turkish validity and reliability study, the scale was reported to have a single-factor structure with a Cronbach's alpha coefficient of 0.81. In the present study, Cronbach's alpha coefficients were 0.79 for the pre-test and 0.80 for the post-test.
Coping Attitudes Assessment Scale | six months
  The scale was originally developed by Carver et al. (1989) and adapted into Turkish by Dicle and Ersanlı (2015). The adapted version consists of 32 items and 5 subscales: Self-Help, Approach, Adaptation, Avoidance-Escape, and Self-Punishment. Items are rated on a four-point Likert-type scale, with higher total scores indicating more effective coping attitudes. In the Turkish validity and reliability study, the overall internal consistency coefficient was reported as 0.97, with Cronbach's alpha values for the subscales ranging from 0.96 to 0.99. In the present study, the overall internal consistency of the scale was 0.78 in the pre-test and 0.81 in the post-test, while Cronbach's alpha values for the subscales ranged between 0.79 and 0.82.

CONTACTS AND LOCATIONS:
Locations (1):
- Buca Seyfi Demirsoy Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No